CLINICAL TRIAL: NCT00837733
Title: Endometrial Local Injury Improves the Pregnancy Rate Among Recurrent Implantation Failure Patients Undergoing IVF/ICSI
Brief Title: Endometrial Local Injury and Implantation Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yazd Research & Clinical Center for Infertility (Other)
Collaborators: Yazd Medical University (Other)
Responsible Party: Department of Obstetrics and Gynecology, Yazd Research & Clinical Center for Infertility
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1551354
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Infertility
Keywords: Endometrial biopsy; IVF/ICSI; Pregnancy outcome; Recurrent implantation failure
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biopsy catheter (Experimental): Biopsy catheter (Pipelle de Cornier, Prodimed, Neuilly-en-Thelle, France
  Interventions: Procedure: Endometrial biopsy

INTERVENTIONS:
Procedure: Endometrial biopsy — Endometrial biopsy was done at luteal phase on the day 21-26 of spontaneous menstrual cycles, when GnRH agonist uses begun. Endometrial samples were taken by a biopsy catheter
  Other Names: biopsy catheter (Pipelle de Cornier, Prodimed, France
Procedure: Endometrial Biopsy — Biopsy catheter
  Other Names: Pipelle de Cornier, Prodimed, Neuilly-en-Thelle, France

SUMMARY:
The purpose of this study is to evaluate the influence of endometrial biopsy on increasing implantation rate in patients with recurrent implantation failures, 93 women with at least two implantation failures were evaluated. In case group endometrial biopsy was obtained from 48 patients in the luteal phase of previous cycle and implantation and clinical pregnancy rate were compared with 45 patients in control group. The results suggest that in vitro fertilization or intracytoplasmic sperm injection after endometrial biopsy increase pregnancy outcome.

DETAILED DESCRIPTION:
In a randomized control trial study, 93 women with at least two implantation failures were evaluated. In case group endometrial biopsy was obtained from 48 patients in the luteal phase of previous cycle and implantation and clinical pregnancy rate were compared with 45 patients in control group.

The implantation rate was determined as 10.9% in biopsy group compared with 3.38% in controls. Clinical pregnancy rate was significantly higher in case group than controls (27.1% and 8.9% respectively

ELIGIBILITY:
Inclusion Criteria:

* women with recurrent implantation failure which was defined as 2-6 cycles unsuccessful of IVF-ET in which more than 10 high grade embryo were transferred

Exclusion Criteria:

* age over than 40 years old
* poor responders to ovarian stimulation

Ages: 15 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Implantation Rate,Chemical pregnancy rate, Clinical pregnancy rate | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Karimzadeh, Professor, Principal Investigator — Research and Clinical Center for Infertility
Locations (1):
- Research and Clinical Center for Infertility, Yazd, Yazd Province, Iran

REFERENCES:
- [Derived] Lensen SF, Armstrong S, Gibreel A, Nastri CO, Raine-Fenning N, Martins WP. Endometrial injury in women undergoing in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Jun 10;6(6):CD009517. doi: 10.1002/14651858.CD009517.pub4. PMID 34110001